CLINICAL TRIAL: NCT02487875
Title: The One Repetition Maximum Test and the Sit-to-stand Test in the Assessment of a Specific Pulmonary Rehabilitation Program on Peripheral Muscle Strength in COPD Patients
Brief Title: Sit-to-stand and Peripheral Muscle Strength in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maugeri Foundation (Other)
Responsible Party: Principal Investigator, Andrea Zanini, MD, Maugeri Foundation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Maugeri1
Record Dates: First submitted 2015-06-25; First posted 2015-07-02 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: COPD
Keywords: Sit-to-stand test; Muscle strength; Pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- COPD patients -study group (Experimental): COPD inpatients GOLD2-4, in stable conditions,hospitalized to follow a pulmonary rehabilitation programme. The study group performs in addition to the standard programme, also a peripheric muscle strength training
  Interventions: Other: rehabilitation
- COPD patients -control group (Active Comparator): COPD inpatients GOLD2-4, in stable conditions,hospitalized to follow a pulmonary rehabilitation programme
  Interventions: Other: rehabilitation

INTERVENTIONS:
Other: rehabilitation

SUMMARY:
Background: Individuals with COPD may present reduced peripheral muscle strength, which leads to impaired mobility. Comprehensive pulmonary rehabilitation (PR) should include strength training, in particular to lower limbs. Furthermore, simple tools for the assessment of lower extremity muscles' performance are required. Objectives: To assess the muscle strength of COPD patients by the sit-to-stand test (STST) as compared to the one-repetition maximum (1-RM), considered as the gold standard in non-laboratory situations, and to evaluate the responsiveness of STST to a PR program with specific strength training (SPR), compared to usual PR program (UPR). Methods: 60 moderate-to-severe COPD inpatients were randomly included into either the SPR or into the UPR. 30-sec STST, 1-min STST, 1-RM and 6MWT were assessed before and after PRs.

DETAILED DESCRIPTION:
Background: Individuals with COPD may present reduced peripheral muscle strength, which leads to impaired mobility. Comprehensive pulmonary rehabilitation (PR) should include strength training, in particular to lower limbs. Furthermore, simple tools for the assessment of lower extremity muscles' performance are required. Objectives: To assess the muscle strength of COPD patients by the sit-to-stand test (STST) as compared to the one-repetition maximum (1-RM), considered as the gold standard in non-laboratory situations, and to evaluate the responsiveness of STST to a PR program with specific strength training (SPR), compared to usual PR program (UPR). Methods: 60 moderate-to-severe COPD inpatients were randomly included into either the SPR or into the UPR. 30-sec STST, 1-min STST, 1-RM and 6MWT were assessed before and after PRs.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis for COPD according to the GOLD criteria.
* no exacerbations over the previous four weeks
* completing PR program
* smoking history ≥10 pack years
* regular treatment with inhaled bronchodilators and inhaled steroids

Exclusion Criteria:

* any unstable medical condition
* Contraindications for participation in the PR program included musculoskeletal disorders, malignant diseases, unstable cardiac condition, and lack of adherence to the program

Ages: 18 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
evaluate the lower limbs' muscle strength by two STSTs (30-sec and 1-min), as compared to the 1-RM in patients with clinically stable COPD, both at baseline and after a PR with specific lower limbs' muscle strength training (SPR). | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Maugeri di Tradate, Tradate, VA, Italy